CLINICAL TRIAL: NCT00754312
Title: A Phase I, Multicenter, Open Label Study on the Effects of SNDX-275 on Expression of Biomarkers in Subjects With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SNDX-275-0302
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ER positive
  Interventions: Drug: SNDX-275
- 2 (Experimental): ER negative and/or PR negative histology
  Interventions: Drug: SNDX-275
- 3 (Experimental): triple negative histology (for ER, PR, HER-2)
  Interventions: Drug: SNDX-275

INTERVENTIONS:
Drug: SNDX-275

SUMMARY:
The primary objective of the study is to evaluate changes in the expression of targeted biomarkers in invasive breast cancer tissue before and after SNDX-275 administration.

ELIGIBILITY:
Inclusion criteria:

* Is scheduled for breast biopsy due to a suspicious mass palpable or ≥1 cm on mammogram
* Must be able to receive two doses of study medication 7 days apart prior to surgery
* Has histologically confirmed invasive breast cancer with ER positive, ER and/or PR negative histology or triple negative (for ER, PR, HER-2) histology
* Has an ECOG performance status ≤ 2
* Has no clinically significant laboratory or cardiac abnormalities
* Has a negative serum pregnancy test at Screening as is either post menopausal, sterile or willing to use an approved method of contraception.
* Is able to swallow and retain oral medication

Exclusion criteria:

* Has a concomitant medical condition that precludes adequate study treatment compliance or assessment, such as: a. Bleeding disorders that would increase risks of additional core biopsy for biomarkers b. Morbid obesity
* Is currently receiving treatment with a medication on the prohibited medication list
* Has allergy to benzamides or inactive components of study drug
* Is participating in another clinical trial or has received another investigational agent within 30 days prior to informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02-28 (Actual); Study Completion 2009-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluate changes in the expression of targeted biomarkers in invasive breast cancer tissue before and after SNDX-275 administration | 14 days

SECONDARY OUTCOMES:
Evaluate changes in gene and/or protein expression of exploratory biomarkers in invasive breast cancer tissue before and after SNDX-275 administration, as tissue sample permits. | 14 days
Evaluate safety and tolerability of SNDX-275 as measured by adverse events and changes in laboratory safety parameters | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Monet Bowling, MD, Principal Investigator — Indiana University; Andrew Baildam, MD, Study Chair — Christie Hospital, UK
Locations (1):
- Monet Bowling, MD, Indianapolis, Indiana, United States